CLINICAL TRIAL: NCT05961163
Title: Chronical Illness-related Limitations of the Ability to Cope With Rising Temperatures: an Observational Study (CLIMATE)
Brief Title: Chronical Illness-related Limitations of the Ability to Cope With Rising Temperatures: an Observational Study
Acronym: CLIMATE
Status: Terminated | Type: Observational
Why Stopped: Terminated due to an unusually cold and rainy summer. E.g. in Hamburg the average temperature between 16 July and 15 August 2023 was below 17°C. Collected data will be used to pilot study design and questionnaire. We plan to repeat the study in 2024.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: IPA-2023-01
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Disease; Myocardial Infarction; Heart Failure; Arrhythmias, Cardiac; Peripheral Artery Disease; Stroke; Ischemic Attack, Transient; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency; Depressive Disorder; Anxiety Disorders; Schizophrenia; Peripheral Nervous System Diseases
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction; Heart Failure; Arrhythmias, Cardiac; Peripheral Arterial Disease; Stroke; Ischemic Attack, Transient; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency; Depressive Disorder; Anxiety Disorders; Schizophrenia; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CLIMATE Observational Study examines to what extent chronically ill patients experience adverse health effects because of heat and whether the patients' specific efforts, somatosensory amplification, self-efficacy, health literacy and commitment to the GP, degree of urbanisation of the patients' administration district and characteristics of the patients' neighborhood are associated with these effects.

DETAILED DESCRIPTION:
The CLIMATE Observational Study aims to analyse to what extent chronically ill patients experience adverse health effects because of heat and whether the patients' specific efforts, self-efficacy, or other factors are associated with these effects. This cohort study is based on an online survey of patients with chronic illness who are recruited in GP practices across all regions of Germany. After the baseline assessment, participants fill out symptom diaries on one specific day of observation per week over a maximum period of 12 weeks. The specific days of observation within the time frame between 29 July and 8 September are selected based on the maximum temperature that can be expected within the respective weeks. The weather forecast will be checked every Friday. If, in the upcoming 4 days, the maximum temperature is expected to exceed 30°C, the warmest day in this time frame will be chosen. Otherwise, the weather forecast will be checked again on Tuesday to choose the warmest of the remaining days of the week. The specific days of observation within the time frame between 9 September and 27 October are randomly selected. On each day of observation, patients are notified by email at 6 pm.

Baseline assessment includes socio-demographic data, health-related quality of life, efforts against adverse effects of heat, somatosensory amplification, self-efficacy, health literacy and commitment to the GP. Local data on temperatures and humidity will be assessed by the measurement stations of Germany's National Meteorological Service. Degree of urbanisation of administration districts is provided by the German Federal Institute for Research on Building, Urban Affairs and Spatial Development. Additionally, small scale data on population density, number of one-person households, unemployment rates and other neighbourhood characteristics are provided by the German Statistical Offices. Data will be analyzed by multivariable, multilevel regression analyses adjusted for possible confounders and random effects on the administration district and practice within administration district level.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older
* at least one of the following conditions: Coronary Heart Disease; Myocardial Infarction; Heart Failure (NYHA stage II or higher); Cardiac Arrhythmias (treated with medication); Peripheral Artery Disease (Fontaine-Ratschow stage II or higher); Stroke; Transient Ischemic Attack; Diabetes Mellitus (Type 1 or 2 treated with oral medication or insulin); Chronic Obstructive Pulmonary Disease (GOLD stage 2 or higher); Asthma (GINA stage II or higher); Renal Insufficiency (KDIGO stage III or higher), Depressive Disorder (treated with medication); Anxiety Disorders (treated with medication), Schizophrenia (treated with medication); Peripheral Nervous System Diseases (with regularly or persistently occurring symptoms).

Exclusion Criteria:

* no capacity to consent
* severe visual impairment
* insufficient German language skills
* not able to use internet browser (eg, lack of hardware)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is located in different sites in Germany. Patients from approximately 50 GP practices will be included. In each practice, eligible patients receive a flyer including a QR-Code and a short link to register for the online study. After documenting informed consent within the application, patients fill out the baseline questionnaire and receive invitations for twelve subsequent assessments of symptoms by email. The investigators estimated that approximately 1500 patients will be contacted. From experience with similar studies the investigators anticipated a response rate of 40% (=600 patients).
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Composite index of nausea, vomiting, tiredness/fatigue, vertigo, circulation problems/syncopes, muscle cramps, headache, extrasystoles, palpitations, edemas, shortness of breath, depressive mood, anxiety, mental confusion | Once per week between 29 July - 27 October 2023
  The severity in each symptom category is defined by the degree of limitations in usual activities. The composite index expresses the highest severity within any symptom category.

SECONDARY OUTCOMES:
Self-rated health | Once per week between 29 July - 27 October 2023
  Measured by visual analogue scale
Use of medical services | Once per week between 29 July - 27 October 2023
  As part of the symptom diary, we will also assess the use of medical services at the specific day of observation (i.e., ambulant care, emergency care, hospital admission)
Reasons for drop out (eg, bad health condition, hospital admission, death) | Once after 27 October 2023
  We will ask participants at baseline for permission to contact any confidential contact in case they drop out from the study

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Schäfer, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Martin Scherer, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will be available from the corresponding authors of study publications upon reasonable request.

REFERENCES:
- [Derived] Jordan A, Nothacker J, Paucke V, Hager KH, Hueber S, Karimzadeh A, Kotter T, Loffler C, Muller BS, Tajdar D, Luhmann D, Scherer M, Schafer I. Association Between Self-Reported Protective Behavior and Heat-Associated Health Complaints Among Patients With Chronic Diseases in Primary Care: Results of the CLIMATE Pilot Cohort Study. JMIR Public Health Surveill. 2024 Nov 4;10:e58711. doi: 10.2196/58711. PMID 39496153